CLINICAL TRIAL: NCT04321616
Title: The (Norwegian) NOR Solidarity Multicenter Trial on the Efficacy of Different Anti-viral Drugs in SARS-CoV-2 Infected Patients
Brief Title: The Efficacy of Different Anti-viral Drugs in COVID 19 Infected Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Barratt-Due, Principal investigator, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118684
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV Infection; COVID 19; Acute Respiratory Distress Syndrome ARDS
Keywords: Effect of drugs; Adverse effects of drugs; SARS-CoV clearance; Duration of artificial ventilation; Duration of intensive care stay; Duration of hospital stay
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Hydroxychloroquine; remdesivir; Standard of Care

STUDY DESIGN:
Intervention Model Description: An open randomized adaptive controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine (Active Comparator)
  Interventions: Drug: Remdesivir; Other: (Standard of Care) SoC
- Remdesivir (Active Comparator)
  Interventions: Drug: Hydroxychloroquine; Other: (Standard of Care) SoC
- Control group - SoC (Active Comparator)
  Interventions: Drug: Hydroxychloroquine; Drug: Remdesivir

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine will be given orally (in the ICU in gastrointestinal tubes) with 800 mg x 2 loading dose followed by 400 mg x 2 every day for a total of 10 days.
  Arms: Control group - SoC; Remdesivir
Drug: Remdesivir — Remdesivir will be given intravenously 100 mg daily for the duration of the hospitalization and up to 10 days total course. A loading dose of 200 mg at inclusion will be given.
  Arms: Control group - SoC; Hydroxychloroquine
Other: (Standard of Care) SoC — The standard of care will be supplied to all patients not receiving a drug intervention.
  Arms: Hydroxychloroquine; Remdesivir

SUMMARY:
The (World Health Organization) WHO NOR- (Coronavirus infectious disease) COVID 19 study is a multi-centre, adaptive, randomized, open clinical trial to evaluate the safety and efficacy of hydroxychloroquine, remdesivir and standard of care in hospitalized adult patients diagnosed with COVID-19. This trial will follow the core WHO protocol but has additional efficacy, safety and explorative endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, 18 years and above
2. Confirmed SARS-2-CoV-2 infection by PCR
3. Admitted to the hospital ward or the ICU
4. Subjects (or legally authorized representative) provides written informed consent prior to initiation of the study

Exclusion Criteria:

1. Severe co-morbidity with life expectancy <3 months according to investigators assessment
2. (Aspartate Transaminase/ Alanine Aminotransferase) ASAT/ALAT > 5 times the upper limit of normal
3. Acute co-morbidity within 7 days before inclusion such as myocardial infarction
4. Known intolerance to the available study drugs
5. Pregnancy, possible pregnancy or breast feeding
6. Any reason why, in the opinion of the investigators, the patient should not participate
7. Subject participates in a potentially confounding drug or device trial during the course of the study
8. Prolonged QT interval (>450 ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 3 weeks
  All cause in-hospital mortality

SECONDARY OUTCOMES:
Occurrence and duration of mechanical ventilation | 3 weeks
Occurrence and duration of intensive care unit (ICU) treatment | 3 weeks
Duration of hospital admittance | 1 month
28 Day mortality | 3 weeks
Viral clearance as assessed by SARS-CoV-2 PCR in peripheral blood and nasopharyngeal airway speciemen | 3 weeks
Occurrence of co-infections | 3 weeks
Occurrence of organ dysfunction | 3 months

OTHER OUTCOMES:
Inflammatory and anti-inflammatory mediators as assessed in serum and plasma | Throughout hospitalization
Markers of extracellular matrix remodeling | Throughout hospitalization and 3 months after remission
Markers of endothelial activation | Throughout hospitalization
Markers of platelet activation | Throughout hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aukrust, MD, Professor, Study Chair — Oslo University Hospital; Andreas Barratt-Due, MD, PhD, Principal Investigator — Oslo University Hospital; Trine Kåsine, MD, Principal Investigator — Oslo University Hospital; Katerina Nezvalova-Henriksen, Pharm D, PhD, Principal Investigator — Oslo Hospital Pharmacies; Anne Margarita Dyrhol Riise, MD, Professor, Principal Investigator — Oslo University Hospital; Marius Trøseid, MD, PhD, Principal Investigator — Oslo University Hospital; Inge Christoffer Olsen, PhD, Principal Investigator — NorCRIN
Locations (1):
- Andreas Barratt-Due, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
All patients included in this study will automatically be included in the WHO COVID 19 protocol
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will end according the requirements to WHO
Access Criteria: WHO COVID 19 investigators

REFERENCES:
- [Derived] Patrick-Brown TDJH, Barratt-Due A, Troseid M, Dyrhol-Riise AM, Nezvalova-Henriksen K, Kasine T, Aukrust P, Olsen IC; NOR Solidarity consortium. The effects of remdesivir on long-term symptoms in patients hospitalised for COVID-19: a pre-specified exploratory analysis. Commun Med (Lond). 2024 Nov 12;4(1):231. doi: 10.1038/s43856-024-00650-4. PMID 39533001
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Tveita A, Murphy SL, Holter JC, Kildal AB, Michelsen AE, Lerum TV, Kaarbo M, Heggelund L, Holten AR, Finbraten AK, Muller KE, Mathiessen A, Boe S, Fevang B, Granerud BK, Tonby K, Lind A, Dudman SG, Henriksen KN, Muller F, Skjonsberg OH, Troseid M, Barratt-Due A, Dyrhol-Riise AM, Aukrust P, Halvorsen B, Dahl TB, Ueland T; NOR-SOLIDARITY Consortium and the Norwegian SARS-CoV-2 Study Group Investigators. High Circulating Levels of the Homeostatic Chemokines CCL19 and CCL21 Predict Mortality and Disease Severity in COVID-19. J Infect Dis. 2022 Dec 13;226(12):2150-2160. doi: 10.1093/infdis/jiac313. PMID 35876699
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Derived] Barratt-Due A, Olsen IC, Nezvalova-Henriksen K, Kasine T, Lund-Johansen F, Hoel H, Holten AR, Tveita A, Mathiessen A, Haugli M, Eiken R, Kildal AB, Berg A, Johannessen A, Heggelund L, Dahl TB, Skara KH, Mielnik P, Le LAK, Thoresen L, Ernst G, Hoff DAL, Skudal H, Kittang BR, Olsen RB, Tholin B, Ystrom CM, Skei NV, Tran T, Dudman S, Andersen JT, Hannula R, Dalgard O, Finbraten AK, Tonby K, Blomberg B, Aballi S, Fladeby C, Steffensen A, Muller F, Dyrhol-Riise AM, Troseid M, Aukrust P; NOR-Solidarity trial. Evaluation of the Effects of Remdesivir and Hydroxychloroquine on Viral Clearance in COVID-19 : A Randomized Trial. Ann Intern Med. 2021 Sep;174(9):1261-1269. doi: 10.7326/M21-0653. Epub 2021 Jul 13. PMID 34251903